CLINICAL TRIAL: NCT03282500
Title: Advances in Treatment: Examining the Effectiveness of a Behavioral Intervention.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kessler Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R-858-14
Record Dates: First submitted 2017-09-12; First posted 2017-09-14 (Actual); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Psychosocial Problems
MeSH Terms: interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to either the experimental condition or the active control condition.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The participants and outcomes assessor are blind to the assigned condition.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness Based Cognitive Therapy (Experimental): In the experimental condition, participants will receive 12 sessions including the instruction of mindfulness skills and cognitive behavioral therapy.
  Interventions: Behavioral: Mindfulness Based Cognitive Therapy
- Psychoeducation on brain injury and treatment (No Intervention): In the control condition, participants will receive 12 sessions on the psychoeducation of brain injuries, outcomes, treatment, and support.

INTERVENTIONS:
Behavioral: Mindfulness Based Cognitive Therapy — The Mindfulness Based Cognitive Therapy (MBCT) intervention promotes self-regulation of emotions and behaviors within an accepting and non-judgmental therapeutic environment. During this interactive, multisensory program, participants will learn strategies to help manage their emotions and thoughts and help them to develop greater insight into the influence these experiences have on their behaviors. Participants will engage in brief at home exercises to enhance their learning of these new skills.
  Arms: Mindfulness Based Cognitive Therapy

SUMMARY:
The purpose of this research is to investigate the influence a mindfulness based cognitive therapy (MBCT) intervention will have on internalizing and externalizing problems in children and adolescents that have suffered a Traumatic Brain Injury (TBI). MBCT is a manualized intervention developed to increase social-emotional resiliency through mindful attention. Internalizing problems refer to a set of symptoms in which a person over-controls their emotions and results in social withdrawal, feelings of worthlessness, depression, and anxiety (Bloom et al., 2001). In contrast, externalizing problems refer to an under-control of emotions which results in conduct problems, impulsive behavior, and aggression. Social and emotional difficulties are prominent consequences of childhood TBI. Left untreated or undertreated, these problems often persist into adulthood, producing a wide range of challenges adapting in personal and vocational domains. At present, there are minimal non-pharmacological therapeutic approaches that effectively treat psychosocial deficits unique to TBI. Developing innovative, evidence based methods is essential in helping children recover from the injury.

DETAILED DESCRIPTION:
Traumatic Brain Injury (TBI) represents a significant, adverse life event. Among the estimated 634,000 pediatric TBI cases occurring annually in the United States (Langlois, Rutlan-Brown, & Thomas, 2006), some reports suggest that approximately 50% of these children and adolescents will develop emotional and behavioral problems. For example, pediatric TBI is associated with negative psychosocial health outcomes including symptoms of internalizing such as depression, (Bloom et al., 2001; Fann, Hart, & Schomer, 2009), withdrawal, and anxiety, and symptoms of externalizing such as impulsivity and aggression (Iversion, 2005; Cole et al., 2008). These maladaptive symptoms are typically correlated with problems in interpersonal relationships and overall social adjustment, contributing to further detriment to social and emotional development (Ganesalingam et al., 2011).

Despite these statistics, our understanding of how to best treat problematic psychosocial sequelae that follow pediatric TBI is largely uncertain and remains an understudied area in the literature. Indeed, relatively few empirically rigorous studies have been conducted examining effective treatment methods targeting internalizing and externalizing symptoms among youth with a TBI; yet, this is an essential area of study that needs to be a priority in research efforts (Semrud-Clikeman, 2010).

Given the beneficial outcomes found with other pediatric populations, it is expected that the MBCT intervention would have a similar, positive impact on adjustment among children and adolescents post TBI. Problems in impulsivity, emotional lability, and anxiety are experienced by many children and adolescents with a TBI, suggesting that a MBCT intervention, which focuses on improving attention, regulatory processes, and reducing stress, would be particularly advantageous for this population.

Youth that meet the inclusion / exclusion criteria will be randomly assigned to either the control group (arts and crafts activities group) or the MBCT experimental condition. The treatments will be 75 minute, weekly sessions for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Moderate or severe Traumatic Brain Injury (TBI)
* TBI occurred at least 6 months prior
* Age at enrollment: 9 to 17 years.
* Elevated internalizing or externalizing symptoms

Exclusion Criteria:

* Substantial impairment in language ability

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Estimated)
Dates: Start 2015-06 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Internalizing Symptoms | 8 weeks
  We will examine the extent to which participants that have completed the experimental condition demonstrate a decrease in Internalizing symptoms (i.e., over-controlling emotions resulting in symptoms of depression and anxiety).
Externalizing Symptoms | 8 weeks
  We will examine the extent to which participants that have completed the experimental condition demonstrate a decrease in Externalizing symptoms (i.e., under-controlling emotions resulting in symptoms of impulsivity, hyperactivity, and aggression).
Adaptive Functioning | 8 weeks
  We will examine the extent to which participants that have completed the experimental condition demonstrate an increase in adaptive functioning (i.e., resilience, social skills, leadership, activities of daily living, and functional communication).

SECONDARY OUTCOMES:
Attention | 8 weeks
  We will examine the extent to which participants that have completed the experimental condition demonstrate a decrease in attention problems.

CONTACTS AND LOCATIONS:
Locations (1):
- Kessler Foundation, East Hanover, New Jersey, United States

REFERENCES:
- [Background] Bloom DR, Levin HS, Ewing-Cobbs L, Saunders AE, Song J, Fletcher JM, Kowatch RA. Lifetime and novel psychiatric disorders after pediatric traumatic brain injury. J Am Acad Child Adolesc Psychiatry. 2001 May;40(5):572-9. doi: 10.1097/00004583-200105000-00017. PMID 11349702
- [Background] Fann JR, Hart T, Schomer KG. Treatment for depression after traumatic brain injury: a systematic review. J Neurotrauma. 2009 Dec;26(12):2383-402. doi: 10.1089/neu.2009.1091. PMID 19698070
- [Background] Cole WR, Gerring JP, Gray RM, Vasa RA, Salorio CF, Grados M, Christensen JR, Slomine BS. Prevalence of aggressive behaviour after severe paediatric traumatic brain injury. Brain Inj. 2008 Nov;22(12):932-9. doi: 10.1080/02699050802454808. PMID 19005885
- [Background] Ganesalingam K, Yeates KO, Taylor HG, Walz NC, Stancin T, Wade S. Executive functions and social competence in young children 6 months following traumatic brain injury. Neuropsychology. 2011 Jul;25(4):466-76. doi: 10.1037/a0022768. PMID 21463038
- [Background] Langlois J, Rutland-Brown W, Thomas K. Traumatic Brain Injury in the United States: Emergency Department Visits, Hospitalizations, and Deaths. Atlanta, GA: Centers for Disease Control and Prevention, National Center for Injury Prevention and Control, 2006.
- [Background] Semrud-Clikeman M. Pediatric traumatic brain injury: rehabilitation and transition to home and school. Appl Neuropsychol. 2010 Apr;17(2):116-22. doi: 10.1080/09084281003708985. PMID 20467952
- [Background] Iverson GL. Outcome from mild traumatic brain injury. Curr Opin Psychiatry. 2005 May;18(3):301-17. doi: 10.1097/01.yco.0000165601.29047.ae. PMID 16639155